CLINICAL TRIAL: NCT04753658
Title: REAL WORLD DATA COLLECTION AMONG PEDIATRIC NEUROBLASTOMA PATIENTS TREATED WITH LORLATINIB THROUGH EXPANDED ACCESS PROGRAM
Brief Title: Real World Data Collection Pediatric Neuroblastoma Treated With Lorlatinib
Status: Terminated | Type: Observational
Why Stopped: The study was prematurely discontinued due to operational implementation challenges and insufficient collection of key data due to varied data accessibility across global study sites.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7461036
Record Dates: First submitted 2021-02-08; First posted 2021-02-15 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-05

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — lorlatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- Pediatric Neuroblastoma Patients Treated with Lorlatinib
  Interventions: Drug: lorlatinib

INTERVENTIONS:
Drug: lorlatinib — Oral

SUMMARY:
The overall goal of this real-world data collection is to assess demographic, clinical characteristics and real-world effectiveness of pediatric neuroblastoma patients treated with lorlatinib through the expanded access program.

ELIGIBILITY:
Inclusion Criteria:

* Patient receives lorlatinib through Pfizer's expanded access program for treatment of ALK+ neuroblastoma.
* HCP documentation of at least one tumor assessment of response after patient has had at least one dose of lorlatinib
* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Any patient who does not meet any of the inclusion criteria defined in the previous section.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 50 pediatric patients with ALK-aberrant neuroblastoma being treated with lorlatinib as part of expanded access program will be included.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States
- Australia (2):
  - Westmead Hospital, Westmead, New South Wales
  - ST0683AU - Chris O'Brien Lifehouse, Camperdown, New South Wales, 2050 Australia
- Starship Blood and Cancer Centre, Auckland, New Zealand
- Instituto Portugues de Oncologia de Lisboa, Lisbon, Portugal
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam
  - Samsung Medical Center, Seoul
- Sweden (4):
  - Queen Silvia Children's Hospital, Gothenburg
  - HRH Crown Princess Victoria's Children and Youth Hospital, Linköping
  - Karolinska Institutet, Stockholm
  - Norrland University Hospital, Umeå

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7461036

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with anaplastic lymphoma kinase (ALK)-aberrant neuroblastoma who initiated treatment with lorlatinib as part of expanded access program were included in this non-interventional study. Data was collected using the data collection tool (DCT).
Groups:
- Lorlatinib: Participants with ALK-aberrant neuroblastoma who initiated treatment with lorlatinib as part of an expanded access program were included. Data was collected on a continual basis until discontinuation of treatment with lorlatinib, death, loss to follow-up or end of study, whichever occurred first.
Period: Overall Study
Arm/Group | Lorlatinib
Started | 15
Completed | 0
Not Completed | 15
Not completed — Progressive disease | 7
Not completed — Other | 7
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All participants for whom data was collected using the data collection tool and observed in this study were included in the analysis.
Arm/Group | Lorlatinib
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.23 (11.553)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants According to Tumor Response of Primary Tumor (Soft Tissue)
Description: Tumor response was collected by the data collection tool (DCT) and responses included complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD). As per International Neuroblastoma Response Criteria (INRC): CR=<10 millimeter (mm) residual soft tissue at primary site and complete resolution of metaiodobenzylguanidine (MIBG) or [18F] fluorodeoxyglucose (FDG)/positron emission tomography (PET) uptake (for MIBG-nonavid tumors) at primary site; PR: >=30% decrease in longest diameter (LD) of primary site & MIBG or FDG-PET uptake at primary site stable, improved, or resolved; SD: neither sufficient shrinkage for PR nor sufficient increase for PD at the primary site. PD greater than 20% increase in longest diameter taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study) and minimum absolute increase of 5 mm in longest dimension. One participant may have more than one tumor response.
Time Frame: From start of lorlatinib treatment until CR, PR, SD or PD, up to maximum of 36.2 months of treatment (data was retrieved and evaluated retrospectively during approximately 18 months of this study)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib
Number analyzed (Participants) | 15
Participants
  CR | 3
  PR | 3
  SD | 5
  PD | 2
  Missing | 7

2. Primary Outcome: Number of Participants According to Tumor Response of Soft Tissue Metastasis and Bone Metastasis
Description: Tumor response collected by DCT.Response included CR=resolution of all sites of disease; PR:>=30% decrease in sum of diameter of non-primary (NP) target lesion (TL) compared to baseline, non-target (NT) lesion may be stable/small in size, no new lesion,>=50% reduced MIBG absolute(abs) bone score (BS) (relative MIBG BS>=0.1 to <=0.5)/>=50% reduced number of FDG-PET avid bone lesion; PD:new soft tissue lesion (STL) detected by computed tomography (CT)/magnetic resonance imaging (MRI) that's MIBG avid/FDG-PET avid, new STL on anatomic imaging, biopsied, confirmed as neuroblastoma(NB)/ganglioneuroblastoma(GNB),new bone site:MIBG avid/FDG-PET avid (for MIBG non-avid tumor) with CT/MRI finding consistent with tumor/confirmed histologically as NB/GNB; >20% increase in LD as reference smallest sum on study,minimum abs. increase of 5mm in sum of diameter of target STL; SD:No sufficient (suff) shrinkage for PR/suff increase for PD of NP lesion.One participant may have more than 1 tumor response
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib
Number analyzed (Participants) | 15
Participants
  CR | 5
  PR | 5
  SD | 5
  PD | 7
  Missing | 2

3. Primary Outcome: Number of Participants According to Bone Marrow Response
Description: Bone marrow response was collected by the DCT and responses included CR, PR, minimal disease (MD) and SD. As per INRC, CR= bone marrow with no tumor infiltration upon reassessment, independent of baseline tumor involvement; PD= bone marrow without tumor infiltration that became > 5% tumor infiltration upon reassessment; or bone marrow with tumor infiltration that increased by > 2 fold and had > 20% tumor infiltration upon reassessment; MD= Bone marrow with less than or equal to (<=) 5% tumor infiltration and remained > 0 to <= 5% tumor infiltration upon reassessment; or bone marrow with no tumor infiltration that became <= 5% tumor infiltration upon reassessment; or bone marrow with >20% tumor infiltration that had > 0 to <= 5% tumor infiltration upon reassessment and SD= bone marrow with tumor infiltration that remained positive with > 5% tumor infiltration upon reassessment but did not meet CR, MD or PD criteria.
Time Frame: From start of lorlatinib treatment until CR, PR, MD or SD, up to maximum of 36.2 months of treatment (data was retrieved and evaluated retrospectively during approximately 18 months of this study)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib
Number analyzed (Participants) | 15
Participants
  CR | 2
  PR | 0
  MD | 1
  SD | 0
  Missing | 12

4. Primary Outcome: Number of Participants According to Health Care Professional (HCP) Reported Objective Response
Description: Objective response was collected by the DCT and comprised of responses in 3 components based on INRC: primary tumor, soft tissue and bone metastases and bone marrow, CR=All components met criteria for CR; PR=PR in at least one component and all other components are either CR, MD (bone marrow), PR (soft tissue or bone), or not involved (NI); no component with PD; Minor response (MR) = PR or CR in at least one component but at least one other component; no component with PD; SD= SD in one component with no better than SD or NI in any other component; PD=Any component with PD. One participant may have more than one tumor response.
Time Frame: From start of lorlatinib treatment until CR, PR, MR, SD or PD, up to maximum of 36.2 months of treatment (data was retrieved and evaluated retrospectively during approximately 18 months of this study)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib
Number analyzed (Participants) | 15
Participants
  CR | 5
  PR | 7
  MR | 1
  SD | 5
  PD | 9

5. Primary Outcome: Number of Participants According to Derived Objective Response
Description: Derived objective response was derived using rules based on responses in 3 components: primary tumor, soft tissue and bone metastases, and bone marrow. CR=All components met criteria for CR. PR=PR in at least one component and all other components are either CR, MD (in bone marrow), PR (soft tissue or bone) or not involved (NI; no component with PD). MR = PR or CR in at least one component but at least one other component with stable disease; no component with PD. SD = Stable disease in one component with no better than SD or NI in any other component; no component with PD. PD = Any component with PD.
Time Frame: as for outcome 4
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib
Number analyzed (Participants) | 15
Participants
  CR | 2
  PR | 0
  MR | 0
  PD | 8
  Missing | 1
  Not Evaluable | 4

6. Primary Outcome: Number of Participants With Best Overall Response Based on HCP Reported Objective Response
Description: Best overall response based on HCP reported objective response comprised of responses (CR, PR, MR, SD and PD) in 3 components: primary tumor, soft tissue and bone metastases, and bone marrow. CR=All components met criteria for CR. PR=At least one component and all other components are either CR, MD (in bone marrow), PR (soft tissue or bone) or not involved (NI; no component with PD). MR = PR or CR in at least one component but at least one other component with stable disease; no component with PD. SD = It is in one component with no better than SD or NI in any other component PD = Any component with PD. Best overall response taking the HCP reported response observed up to the data cut-off date for a specific milestone.
Time Frame: as for outcome 4
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib
Number analyzed (Participants) | 15
Participants
  CR | 5
  PR | 3
  MR | 1
  SD | 3
  PD | 3

7. Primary Outcome: Number of Participants With Best Overall Response Based on Derived Objective Response
Description: Best overall response based on derived objective response comprised of responses (CR, PR, MR, SD and PD) in 3 components: primary tumor, soft tissue and bone metastases, and bone marrow. CR=All components met criteria for CR. PR=PR in at least one component and all other components are either CR, MD (in bone marrow), PR (soft tissue or bone) or not involved (NI; no component with PD). MR= PR or CR in at least one component but at least one other component with stable disease; no component with PD. SD= Stable disease in one component with no better than SD or NI in any other component; no component with PD. PD= Any component with PD.
Time Frame: as for outcome 4
Population: All participants for whom data was collected using the data collection tool and observed were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib
Number analyzed (Participants) | 15
Participants
  CR | 2
  PD | 8
  Missing | 5

8. Primary Outcome: Overall Response Rate Based on HCP Reported Response
Description: Overall response rate was defined as the percentage of participants with a best overall response of CR or PR. CR=All components (primary tumor, soft tissue and bone metastases, and bone marrow) met criteria for CR. PR=PR in at least one component and all other components are either CR, MD (in bone marrow), PR (soft tissue or bone) or not involved (NI; no component with PD). Two sided 95% confidence interval was based on Clopper Pearson method.
Time Frame: From start of lorlatinib treatment until CR or PR, up to maximum of 36.2 months of treatment (data was retrieved and evaluated retrospectively during approximately 18 months of this study)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lorlatinib
Number analyzed (Participants) | 15
Percentage of participants | 53.3 [26.6 to 78.7]

9. Primary Outcome: Overall Response Rate Based on Derived Response
Description: Overall response rate was defined as the percentage of participants with a best overall response of CR or PR. CR=All components (primary tumor, soft tissue and bone metastases, and bone marrow) met criteria for CR. PR=PR in at least one component and all other components are either CR, MD (in bone marrow), PR (soft tissue or bone) or not involved (NI; no component with PD).
Time Frame: as for outcome 8
Population: All participants for whom data was collected using the data collection tool and observed in this study were included in the analysis. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lorlatinib
Number analyzed (Participants) | 10
Percentage of Participants | 13.3 [1.7 to 40.5]

10. Primary Outcome: Duration of HCP Reported Overall Responses
Description: Duration of HCP reported overall response was derived as (earliest date of disease progression or death minus earliest date of complete or partial response + 1)/30.4. Participants who had not progressed or died were censored at their last assessment date prior to the data cut-off date. CR=All components (primary tumor, soft tissue and bone metastases, and bone marrow) met criteria for CR. PR=PR in at least one component and all other components are either CR, MD (in bone marrow), PR (soft tissue or bone) or not involved. PD=Any component with PD.
Time Frame: From date of CR or PR until earliest date of PD or death or censoring date, up to maximum of 36.2 months of treatment (data was retrieved and evaluated retrospectively during approximately 18 months of this study)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib
Number analyzed (Participants) | 15
Months | 21.7 [2.0 to NA] — The upper limit of its 95% confidence interval was not estimable due to insufficient number of participants with events.

11. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was derived as (date of PD or death [by any cause in the absence of PD] minus date of first dose of lorlatinib plus 1) divided by 30.4. Participants who had not progressed or died were censored at the date of last contact prior to the data cut-off date. PD: new soft tissue lesion (STL) detected by CT/MRI that's MIBG avid/FDG-PET avid, new STL on anatomic imaging, biopsied and confirmed as neuroblastoma (NB)/ganglioneuroblastoma (GNB), new bone site: MIBG avid/FDG-PET avid (for MIBG non-avid tumor) with CT/MRI finding consistent with tumor or confirmed histologically as NB/GNB; >20% increase in LD as reference smallest sum on study (included baseline sum if that was the smallest on study), minimum abs increase of 5mm in sum of diameter of target STL.
Time Frame: From start of lorlatinib treatment until disease progression or death or censoring date, up to maximum of 36.2 months of treatment (data was retrieved and evaluated retrospectively during approximately 18 months of this study)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib
Number analyzed (Participants) | 15
Months | 17.8 [3.7 to NA] — The upper limit of its 95% confidence interval was not estimable due to insufficient number of participants with events.

12. Primary Outcome: Duration of Treatment
Description: Duration of treatment was derived as treatment stop date minus treatment start date plus 1. Participants continuing treatment at the data cut-off date were censored based on the last recorded date when the participant was known to be continuing treatment prior to the data cut-off date.
Time Frame: From start of lorlatinib treatment until treatment stop date or censoring date, up to maximum of 36.2 months of treatment (data was retrieved and evaluated retrospectively during approximately 18 months of this study)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib
Number analyzed (Participants) | 15
Months | 16.2 [3.4 to 24.2]

13. Primary Outcome: Overall Survival
Description: Overall survival was derived as date of death minus treatment start date plus 1. Participants who had not died were censored at the date of last contact prior to the data cut-off date.
Time Frame: From date of first dose of lorlatinib until date of death or censoring date, up to maximum (max) of 36.2 months (M) of treatment (data was retrieved and evaluated retrospectively during approximately (approx.) 18 months of this study)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib
Number analyzed (Participants) | 15
Months | 27.0 [4.8 to NA] — The upper limit of its 95% confidence interval was not estimable due to insufficient number of participants with events.

14. Primary Outcome: Number of Participants Reporting Adverse Events, Treatment-Related Adverse Events, Serious Adverse Events and Treatment-Related Serious-Adverse Events
Description: An AE is any untoward medical occurrence in participants administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. A SAE is any untoward medical occurrence in a participant administered a medicinal or nutritional product at any dose that: resulted in death, was life-threatening, required participant hospitalization or prolongation of hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions) and resulted in congenital anomaly/birth defect. Relatedness to treatment was determined by investigator.
Time Frame: From start of first dose of lorlatinib/date of informed consent(participant treated with lorlatinib) to atleast 28 day after last dose of lorlatinib to max 36.2M of treatment(data was retrieved, evaluated for approx. 18 month)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib
Number analyzed (Participants) | 15
Participants
  AEs | 14
  Treatment related AEs | 14
  Serious AEs | 6
  Serious Treatment related AEs | 3

ADVERSE EVENTS:
Time Frame: From start of first dose of lorlatinib or date of informed consent (for participants being treated with lorlatinib at study start) until at least 28 days following last administration of lorlatinib (maximum treatment duration of 36.2 months), data was retrieved and evaluated retrospectively during approx.18 months of this study
Description: An AE term may be reported as both a serious and non-serious AE but are distinct events. An AE may be serious for 1 participant and non-serious for another participant, or a participant may have experienced both a serious and non-serious episode of the same event.
Arm/Group | Lorlatinib
All-Cause Mortality (participants affected / at risk) | 8/15
Serious Adverse Events (participants affected / at risk) | 6/15
Other Adverse Events (participants affected / at risk) | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lorlatinib (N=15)
Hemiparesis (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Pneumonia (Infections and infestations) | 1
Rhinovirus infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Weight increased (Investigations) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Primary hypogonadism (Endocrine disorders) | 1
Pyrexia (General disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urinary retention (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lorlatinib (N=15)
Blood cholesterol increased (Investigations) | 6
Weight increased (Investigations) | 6
Alanine aminotransferase increased (Investigations) | 3
Blood triglycerides increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Fine motor delay (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Speech disorder developmental (Nervous system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Candida infection (Infections and infestations) | 2
Pyelonephritis (Infections and infestations) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Oedema peripheral (General disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Insomnia (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/58/NCT04753658/Prot_SAP_000.pdf